CLINICAL TRIAL: NCT06076499
Title: A Post-Market Observational Clinical Study to Determine the Long-Term Effectiveness and Safety of the Noctrix NTX100 TOMAC (Tonic Motor Activation) System for the Treatment of Restless Legs Syndrome - The THRIVE Study
Brief Title: A Post-Market Study for Long-Term Effectiveness and Safety of the NTX100 for RLS
Acronym: THRIVE
Status: Active, not recruiting | Type: Observational
Sponsor: Noctrix Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-06
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Restless Legs Syndrome
Keywords: RLS
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: NTX100 — NTX100 Tonic Motor Activation (TOMAC) System - a non-invasive peripheral nerve stimulation device programmed to deliver active stimulation.

SUMMARY:
Multi-center post-market, observational study to assess the long-term effectiveness and safety of the NTX100 TOMAC System for patients with Restless Legs Syndrome.

DETAILED DESCRIPTION:
This study will assess the NTX100 TOMAC System's long-term effectiveness and safety in real-world settings. Using a prospective, observational approach, we'll monitor individuals receiving the system as part of standard care through five study visits, collecting data on clinical outcomes, device performance, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The subject possesses the necessary equipment, internet/phone accessibility, and communication ability to complete electronic questionnaires and respond to electronic communications and phone calls from the research staff throughout the in-home portion of the study.
2. The subject has signed a valid, IRB-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English.
3. Diagnosis of restless legs syndrome.

Exclusion Criteria:

1. The subject is unable or unwilling to comply with study requirements.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults who meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 1 year
  Change from baseline (study entry) in IRLS total score at 1-year.

SECONDARY OUTCOMES:
CGI-I score at 1-year relative to baseline | 1 year
  The 1-year Clinical Global Impression-Improvement (CGI-I) score assesses a patient's overall condition relative to their baseline, indicating treatment effectiveness and change in condition over a year. Scores range from 1 (very much improved) to 7 (very much worse).
PGI-I Score at 1-Year Relative to Baseline | 1 year
  The 1-year Patient Global Impression-Improvement (PGI-I) score assesses the patient's perception of their condition's improvement from baseline, with scores ranging from 1 (very much improved) to 7 (very much worse).
Change from baseline in MOS-II total score at 1-year. | 1-year
  The Medical Outcomes Study 36-Item Short Form Health Survey (MOS-II) measures various aspects of a patient's health-related quality of life. This endpoint assesses the change in the total MOS-II score at the 1-year mark compared to the baseline, and how the treatment impacts overall well-being over the course of a year.
Change from Baseline in Frequency of RLS Symptoms (Number of Days per Week) at 1-Year | 1-year
  This endpoint focuses on Restless Legs Syndrome (RLS) and assesses the change in symptom frequency over a year. It quantifies the reduction in the number of days per week that a patient experiences RLS symptoms, indicating the treatment's effectiveness in managing this condition over time.

OTHER OUTCOMES:
CGI-I responder rate, defined as a CGI-I response of "Very Much Improved" or "Much Improved", at 1-year. | 1-year
  This metric gauges the proportion of patients showing significant improvement after one year of treatment, defined as a "Very Much Improved" or "Much Improved" CGI-I response.
CGI-I improvement rate, defined as the percentage of patients with a CGI-I response of "Very Much Improved", "Much Improved" or "Minimally Improved". | 1-year
  This measure indicates the percentage of patients experiencing positive change due to treatment, encompassing "Very Much Improved," "Much Improved," and "Minimally Improved" CGI-I responses.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Preciado, PhD, Study Director — Noctrix Health, Inc.
Locations (6):
- United States (6):
  - Mark J Buchfuhrer, MD Office, Downey, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - Neurocare, Inc., Newton, Massachusetts
  - Clayton Sleep Institute, St Louis, Missouri
  - Ohio Sleep Medicine and Institute, Dublin, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina

REFERENCES:
- [Background] Buchfuhrer MJ, Baker FC, Singh H, Kolotovska V, Adlou B, Anand H, de Zambotti M, Ismail M, Raghunathan S, Charlesworth JD. Noninvasive neuromodulation reduces symptoms of restless legs syndrome. J Clin Sleep Med. 2021 Aug 1;17(8):1685-1694. doi: 10.5664/jcsm.9404. PMID 33949942
- [Background] Charlesworth JD, Adlou B, Singh H, Buchfuhrer MJ. Bilateral high-frequency noninvasive peroneal nerve stimulation evokes tonic leg muscle activation for sleep-compatible reduction of restless legs syndrome symptoms. J Clin Sleep Med. 2023 Jul 1;19(7):1199-1209. doi: 10.5664/jcsm.10536. PMID 36856064
- [Background] Bogan RK, Roy A, Kram J, Ojile J, Rosenberg R, Hudson JD, Scheuller HS, Winkelman JW, Charlesworth JD. Efficacy and safety of tonic motor activation (TOMAC) for medication-refractory restless legs syndrome: a randomized clinical trial. Sleep. 2023 Oct 11;46(10):zsad190. doi: 10.1093/sleep/zsad190. PMID 37458698
- [Background] Roy A, Ojile J, Kram J, Olin J, Rosenberg R, Hudson JD, Bogan RK, Charlesworth JD. Long-term efficacy and safety of tonic motor activation for treatment of medication-refractory restless legs syndrome: A 24-Week Open-Label Extension Study. Sleep. 2023 Oct 11;46(10):zsad188. doi: 10.1093/sleep/zsad188. PMID 37439365
- See also: Noninvasive neuromodulation reduces symptoms of restless legs syndrome — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8656897/
- See also: Bilateral high-frequency noninvasive peroneal nerve stimulation evokes tonic leg muscle activation for sleep-compatible reduction of restless legs syndrome symptoms — https://pubmed.ncbi.nlm.nih.gov/36856064/